CLINICAL TRIAL: NCT05460195
Title: Sintilimab Combined With Anlotinib for Perioperative Non-small Cell Lung Cancer Based on MRD Evaluation: a Clinical Study
Brief Title: Sintilimab Combined With Anlotinib for Perioperative Non-small Cell Lung Cancer Based on MRD Evaluation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Tianqing Chu, Associate Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChestKS22002
Record Dates: First submitted 2022-07-03; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Non-small Cell Lung Cancer; Minimal Residual Disease; Immunotherapy; Anti-angiogenesis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm, Residual | interventions — anlotinib; Immunotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination therapy group (Experimental): Sintilimab combined with anlotinib
  Interventions: Drug: sintilimab combined with anlotinib
- Single-agent therapy group (Experimental): Sintilimab monotherapy
  Interventions: Drug: sintilimab monotherapy

INTERVENTIONS:
Drug: sintilimab combined with anlotinib — Sintilimab (200mg/time, every 3 weeks) combined with anlotinib (12mg, once daily on day 1 to 14 per cycle) for 2 cycles (42 days). Radical surgery is performed within 4 - 6 weeks treatment. Sintilimab combined with anlotinib therapy repeats every 3 weeks until one year after surgery.
  Other Names: immunotherapy combined with antiangiogenic therapy
  Arms: Combination therapy group
Drug: sintilimab monotherapy — Sintilimab (200mg/time, every 3 weeks) combined with anlotinib (12mg, once daily on day 1 to 14 per cycle) for 2 cycles (42 days). Radical surgery is performed within 4 - 6 weeks treatment. Sintilimab monotherapy repeats every 3 weeks until one year after surgery.
  Other Names: immunotherapy
  Arms: Single-agent therapy group

SUMMARY:
To study the efficacy of sintilimab combined with anlotinib for perioperative non-small cell lung cancer. To explore the clearance effect of sintilimab combined with anlotinib for postoperative adjuvant therapy based on evaluating minimal residual disease.

DETAILED DESCRIPTION:
Patients with resectable non-small cell lung cancer (NSCLC) have a high postoperative recurrence rate. Perioperative treatment, which can improve the resection rate and clear the minimal residual disease, is the main mean of preventing recurrence, including preoperative neoadjuvant and postoperative adjuvant therapies. In recent years, immunotherapy can significantly improve the pathological remission rate and prolong the survival as a perioperative treatment. In addition to single-agent or combined chemotherapy, the exploration of immunotherapy with other therapeutic strategies is still lacking.

In 2018, we originally designed sintilimab combined with anlotinib in the first-line treatment of advanced NSCLC.

This clinical study plans to: ① apply the "de-chemotherapy" model to the perioperative phase of early NSCLC, ② explore sintilimab combined with anlotinib in preoperative neoadjuvant and postoperative adjuvant therapies, ③ explore clearance effect of sintilimab combined with anlotinib for postoperative adjuvant therapy based on evaluating minimal residual disease (MRD), in order to improve the efficacy of perioperative NSCLC and prolong survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cyologically confirmed stage II-IIIa NSCLC patients;
* NSCLC patients with negative driver gene: EGFR wild-type, no ALK fusion mutation, no ROS1 fusion mutation;
* ECOG PS: 0~1;
* Pulmonary function index meets the surgical criteria;
* No previous systemic anti-tumor treatment.

Exclusion Criteria:

* Patients with central cavitary squamous cell carcinoma or investigator-assessed bleeding symptoms or bleeding tendency were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | 2 months
  Residual tumor cells of the surgical specimens were ≤10% based on pathological evaluation.

SECONDARY OUTCOMES:
Complete pathologic response (CPR) | 2 months
  Residual tumor cells of the surgical specimens were 0% based on pathological evaluation.
Event free survival (EFS) | 16 months
  Time from randomization to any of the following: disease progression; new primary NSCLC; death from any cause
Overall survival (OS) | 32 months
  Radiographic assessments were performed when enrolled and every 8 weeks until disease progression after chemotherapy according to RECIST version 1.1. After PD, collect the survival information every 16 weeks until death or withdrawal of study consent.

CONTACTS AND LOCATIONS:
Overall Officials: Tianqing Chu Chu, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China